CLINICAL TRIAL: NCT06599099
Title: Building Mood State Classifiers to Inform Deep Brain Stimulation of Treatment-Resistant Bipolar Depression
Brief Title: Deep Brain Stimulation of Treatment-Resistant Bipolar Depression
Acronym: DBS in TRBD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne Goodman MD (Other)
Collaborators: University of Washington (Other); William Marsh Rice University (Other); Massachusetts General Hospital (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Wayne Goodman MD, Chairman/Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-53761; 1UH3NS136631 (NIH)
Record Dates: First submitted 2024-08-28; First posted 2024-09-19 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Bipolar Depression
Keywords: Treatment Resistant Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: This model will include 10 subjects between the ages of 22 and 64 with severe, TRBD. These subjects will undergo surgery with DBS leads targeting the ventral capsule/ventral striatum (VC/VS) bilaterally to assess the safety and preliminary efficacy of VC/VS DBS. Subjects will undergo behavioral and clinical testing to provide further insight for alleviating and preventing recurrence of depression and emergence of mania.
Who Masked: Participant, Outcomes Assessor
Masking Description: Discontinuation: In all cases, the sequence will be as follows in one-week segments: 100% Active (Sham discontinuation), 75% Active, 50% Active, 25% Active, and 0% Active (stim off). They will be told that DBS will be discontinued at some point during the 4 weeks. The programmer will be unblinded and perform "sham" activation. Relapse is defined as a 25% increase of the MADRS over two consecutive visits compared to discontinuation baseline. Escape criteria will include withdrawing consent or significant clinical deterioration warranting unblinding or reinstatement of treatment. Following exit from the discontinuation period, treatment will recommence as clinically indicated including stimulation resumption or continued observation with device off. A stepwise discontinuation over 4 weeks is intended to mitigate rebound effects, striking a balance between scientific need and subject well-being, with escape criteria allowing us to re-initiate therapy if needed for patient safety.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Medtronic Percept RC System Implantation for TRBD (Experimental): All subjects will receive surgical implantation of Percept RC DBS system
  Interventions: Device: Medtronic Percept RC System
- One Month Blinded Discontinuation Period (Experimental): The investigators will use blinded discontinuation at 12 months rather than sham control to establish evidence that response is dependent on ongoing DBS.
  Interventions: Behavioral: One Month Blinded Discontinuation Period

INTERVENTIONS:
Device: Medtronic Percept RC System — Medtronic Percept RC System includes:
  Percept RC neurostimulator SenSight Directional Lead Kit (with and without marker; 33cm and 42cm lengths) SenSight Directional Lead Kit (with and without marker; 33cm and 42cm lengths) SenSight Extension Kit (with and without marker; 40cm, 60cm, and 95cm lengths) Percept DBS Handset and Communicator Kit (patient programmer) SenSight Extension Tunneler Kit SenSight Burr Hole Device Kit Clinician Programmer Application (application runs on Model CT900 Tablet) Percept RC Recharger Kit Recharge Application Software Clinician Communicator/Telemetry Module
  Other Names: Deep Brain Stimulation System; DBS
  Arms: Medtronic Percept RC System Implantation for TRBD
Behavioral: One Month Blinded Discontinuation Period — The investigators will use blinded discontinuation at 12 months rather than sham control to establish evidence that response is dependent on ongoing DBS. The open-label design allows for personalized optimization of programming settings - a strength of this design as related to our study goals. Although one of the goals of this study is to use neural recordings to inform programming, currently, unblinded programming is needed to maximize response and minimize side effects. Adverse events will be elicited at each study visit using a standardized instrument, the Patient-Rated Inventory of Side Effects (PRISE). In addition to monitoring for adverse events related to surgery and stimulation, the investigators will track quality of life (QOLS), global functioning (SDS), and necessary adjustments of medications. The behavioral changes of the subject based on these scales will provide insight to the intervention levels provided from discontinuing the therapy from the device.
  Arms: One Month Blinded Discontinuation Period

SUMMARY:
This study is only enrolling at Baylor College of Medicine. The other research locations listed serve to support data analysis only.

This research study is to investigate the use of technology called Deep Brain Stimulation (DBS) to potentially improve Treatment-Resistant Bipolar Depression (TRBD) symptoms in patients with severe cases. DBS involves the surgical implantation of leads and electrodes into specific areas of the brain, which are thought to influence the disease. A pack implanted in the chest, called the neurotransmitter, keeps the electrical current coursing to the brain through a wire that connects the neurotransmitter and electrodes. It is believed DBS may restore balance to dysfunctional brain circuitry implicated in TRBD. The goal of this study is to enhance current approaches to DBS targeting in the brain and to use a novel approach to find a better and more reliable system for TRBD treatment.

Its important for participants to understand that this is an investigational study where there could be a lack of effectiveness in improving TRBD symptoms. There may be no directly benefit from taking part in this study.

This study is expected to last 20 months and involves 3 main steps.

1. Medical, psychiatric, and cognitive evaluations.
2. Implantation of a brain stimulation system.
3. Follow up after implantation of device, including programming, recording, and psychiatric testing.

There are risks and benefits to this study which need to be considered when deciding to participate or not. Some of the risks are from surgery, the DBS device and programming, the tests involved, and potential loss of confidentiality, as well as other unknown risks.

Some of the more serious risks involved in this study and the percentage that they occur:

1. Bleeding inside the Brain (1 to 2 percent).
2. Infection from the procedures (3 percent)
3. Seizure caused from the procedures (1.2 percent)

However, the benefit of this study is that it may help relieve or decrease TRBD symptoms. This form of treatment has shown to reduce symptom severity in other cases. This could potentially improve quality of life and activities in daily routines. There is also a potential benefit to society in that the data the investigators will obtain from this study may help increase the understanding of the mechanisms underlying TRBD symptoms, as well as enhanced Deep Brain Stimulation techniques.

Study participation is expected to last 20 months from the time the DBS device is activated and should include approximately 23 visits. These visits also include 8 separate, 24 hour stays at the Menninger NeuroBehvaioral Monitoring Unit (NBU). These 24-hour sessions will occur at multiple points throughout the study (1 week prior to surgery, the week preceding device activation, the week following activation, then after 2 weeks, 4 weeks, 6 months, 9 months, and 12 months). Participants will need to stay locally for the week of the NBU stay (typically Monday through Friday).

Study visits will include clinician administered assessments and questionnaires, subject reported assessments, neuropsychological testing, and mobile behavioral assessments which will occur around 23 visits over the course of 20 months.

DETAILED DESCRIPTION:
This study is only enrolling at Baylor College of Medicine. The other research locations listed serve to support data analysis only.

Enrollment: A subject is considered enrolled upon signing informed consent and deemed eligible to be screened by the investigator. The informed consent process may include discussions with the patients family and referring clinician.

Screening: Potential subjects meeting inclusion/exclusion criteria and willing to participate in the study as demonstrated by signing the informed consent will be enrolled in the study and undergo a screening and baseline visit (Visit 1 and Visit 2) spaced over an approximate 1 month period. Diagnostic and screening ratings are completed, followed by complete medical, neurological and neurosurgical evaluations. Final selection of candidates will be made by consensus of the multi-disciplinary investigator team.

Surgical Procedures: All patients will be implanted with bilateral leads targeting the VC/VS using the investigators previously described robotic DBS workflow. In brief, preoperative high-resolution MRI (3D, T1-weighted with and without contrast) and 3D CT will be obtained and uploaded to the ROSA (Zimmer Biomet) planning station. Images will be merged, and the AC, posterior commissure, and interhemispheric plane will be marked as is routinely done for stereotactic procedures. The investigatorswill plan two trajectories for each hemisphere and use intraoperative awake testing to validate the optimal target. One trajectory will be planned just anterior to AC (VC/VS), the other just posterior (bed nucleus stria terminalis (BNST)). The investigatorshave successfully implemented intraoperative behavioral testing to adjudicate between VC/VS and BNST in patients with treatment resistant OCD. Both trajectories will be planned such that the deepest contact is at the white/gray matter junction (i.e., VC/VS for the anterior trajectory, BNST for the posterior trajectory). The trajectory will follow the coronal contour of the anterior limb of the internal capsule (ALIC).

The investigators will use the postcontrast scan to ensure lack of vessel collision. A stereotactic frame (Leksell model G, Elekta) will be placed under local anesthesia. Under light sedation (to minimize movement), a fluoroscopic CT scan (O-arm 2, Medtronic) will be obtained and merged with the other image sets on the robotic navigation system. Using the frame skull pins as bone fiducials, the robot will be registered to the fixed head, and entry points marked according to preoperative planning. The head will be prepped and draped to allow for awake evaluation of the patient later in the procedure. The fluoroscopic CT will be draped into the field so that an intraoperative scan can be easily acquired. A single burr hole on each side will be drilled. The burr hole will be large enough to accommodate both trajectories.

Intraoperative Behavioral Testing. Lead securing devices will be installed bilaterally, and sedation stopped for intraoperative testing. A cannula (0 mm above target, 192 mm length, Alpha Omega) will be introduced to the first target as usual in DBS surgery. In general, the left VC/VS will be chosen as the first target. In cases in which the BNST is the safer trajectory, this target will be tested first. A DBS lead will be placed, and the cannula withdrawn to expose the contacts. Intraoperative evaluation will be conducted by a psychiatrist (W.K.G.), including a quick monopolar survey of all 4 contacts up to 5 mA. The investigators will ask whether the patient experiences any change in mood, energy, or anxiety while evaluating for positive valence (PV) affect (improved mood, increased energy, and reduced anxiety) on all contacts, and for adverse effects (increased anxiety, worsened mood, or other negative valence (NV) response). If a strong, consistent PV is produced during the monopolar survey, and no side effects are evident, the lead will be secured in that position. If no PV is evident, or if NV is produced, or other side effects are present, the lead will be removed, and the cannula repositioned to the second target. The investigators will then conduct another monopolar review at the second target in the same manner. Following stimulation of the second target, the neurosurgery and psychiatry teams will discuss the results to choose the final location of the lead. The patient will be blinded to stimulation target, amplitude, and side. The DBS system will be activated approximately 2 weeks following surgery during the first programming visit.

NeuroBehavioral Monitoring Unit (NBU). To capture high-density neural data coupled with multimodal measures (including sleep), subjects will spend 24 hours in the NBU - located at The Menninger Clinic's main campus in Houston - at multiple time points in the study:

1. week prior to surgery and week preceding activation, and
2. week following activation, then after 2 weeks, 4 weeks, 6 months, 9 months, and 12 months.

   The total days in NBU per subject is 8. Each of those visits will correspond to a period "in-situ", which will generally be 5 days long (Monday through Friday), including one day in the NBU. These are times when subjects will reside locally due to frequency of assessments or need for high-density recordings in NBU. In general, subjects will be asked to stay locally (in the greater Houston area) for the first 4 weeks following activation. To support recording neural time-domain local field potentials streaming while in the NBU, a Percept clinician programmer will be placed inside the room and configured to stream from the subject's implanted device for the duration of the participant's stay. A research coordinator will be responsible for restarting streaming sessions every eight hours, ensuring the patient's device stays charged, and ensuring the tablet stays connected as the patient moves through common spaces in on the Menninger campus. The clinician programmer tablet will be physically secured such that the subject cannot mistakenly tamper with it. Within the NBU, the subject will be asked to wear the mobile sensing systems (Apple watch, Oura ring, and audioband) to be deployed in the participant's home for sensor performance characterization.

   Multimodal Biobehavioral Measurement. Unlike movement disorders where the effect of stimulation can be acquired near instantaneously during programming, psychological state fluctuations require monitoring over days or weeks which can be best accomplished using wearable systems in naturalistic settings. The Rune patient app collects patient reported events, diary info and wearable data and pushes it up to the cloud (StrivePD portal). The neural data need to be uploaded to the Rune StrivePD web portal for integrating and synching the neural data with the behavioral data. The Percept-RC sensing capabilities will allow the investigators to collect high density neural data in the clinic and NBU, and less dense but chronic neural data collected in parallel with ecological data obtained outside the clinic. Passive and active (e.g., EMA survey pushes) behavioral data will be collected throughout the clinical trial, including baseline before surgery and baseline pre-activation following surgery.

   Weeks -8-0 (Screening and Baseline) The following Clinician-administered assessments will take place: Vital Signs, Structured Interview (SCID-5), SCID-5-PD (Personality Disorders); Montgomery Asberg Rating Scale (MADRS), Global Severity/Change (CGI-S/I), Young Mania Rating Scale (YMRS)56, Suicidality (C-SSRS), Anxiety (HAM-A), Medication Recommendation Tracking Form (MRTF) , Side-Effects (PRISE),;

   The following Subject Reported assessments will take place: Depression (QIDS-SR), Quality of Life Scale (QOLS), Sheehan Disability (SDS), Barratt Impulsiveness Scale (BIS), Altman Self-Rating Mania Scale (ASRM), Insomnia Severity Index (ISI) , Positive and Negative Affect Schedule (PANAS), Morning-Eveningness Questionnaire (MEQ), Internal State Scale (ISS),;

   The following Medical and Laboratory Testing will take place: Physical Exam, Vital Signs, ECG, UA, CMP, CBC, PT/PTT/INR, Hepatitis serology, pregnancy, tox screen; Brain Imaging: 3T: sMRI, DTI; MEG, rsfMRI.

   All blood draws are for clinical purposes ONLY and not research.

   The following Neuropsychological Testing (Neuropsych) will occur: MMSE, HVLT-R*, BVMT-R*, MoCA, TOPF, Weschler Adult Intelligence Scale IV Edition: Digit Span, Coding, Similarities, Information, Visual Puzzles; Trails A & B; WCST-64Rey-Osterrieth Complex Figure, DKEFS lexical and semantic fluency*, STROOP, BDI-II, PSWQ, OCI-R, Millon Behavioral Medicine diagnostic (MBMD) (baseline only) [Alternate forms for follow-up testing];

   The following Behavioral Tasks will occur: Probabilistic Reward Task (PRT) and Immediate Memory Task (IMT) will be given at baseline Mobile biobehavioral measures: (e.g., Rune app ingested data from wearables, peripherals, self-reports). Administer 5-10-minute Ecological Momentary Assessment (EMA) sessions will be triggered starting at baseline and throughout the course of the study. Peripherals and wearables for activity and sleep monitoring will be provided for continuous use.

   Neurobehavioral Unit: Will be "in-situ" (staying locally) during much of this time and spend one 24-hour period in in a clinical monitoring environment) for highdensity streaming coupled with multi-modal behavioral measures including computer vision for affect and activity analysis, speech analysis, peripherals and wearables for activity and sleep. Polysomnography at baseline overnight stay at NBU to conduct baseline sleep study for validation of concurrent and subsequent Oura Ring sleep monitoring.

   (This will be NBU visit 1 of 8)

   DBS SURGERY VISIT: CT scans will be performed prior to, during and after surgery. The DBS System Implantation of bilateral VC/VS current steering electrodes.

   Week 1-2: Following one week recovery, seen for repeat baseline assessments pre-DBS activation. These include:

   Clinician-administered: Vital Signs, MADRS, CGIS, YMRS, C-SSRS,HAM-A, MRTF, PRISE, Subject Reported: QIDS-SR, QOLS, SDS, BIS, ASRM, PANAS, MEQ, ISS. Medical and Laboratory Testing: Repeat MEG, rsfMRI.

   Neuropsychological Testing (Neuropsych): Repeat the neuropsych battery defined in the screening/baseline period. Behavioral Tasks: PRT, and IMT.

   Mobile Biobehavioral measures: ongoing data collection through continuous use of wearable sensors, peripherals, and EMA.

   NeuroBehavioral Unit: two 24-hour periods in NBU. (This will include NBU visit 2 of 8)

   Week 2 following surgery: Following two week recovery, subject will be seen for baseline assessments and system activation of theDBS device.

   Repeat Assessments:

   Clinician-administered: Vital Signs, MADRS, CGIS, YMRS, C-SSRS, HAM-A, MRTF, PRISE,

   Subject Reported: QIDS-SR, QOLS, SDS, BIS, ASRM, PANAS, MEQ, ISS.

   Neuropsychological Testing (Neuropsych): Repeat the neuropsych battery defined in the screening/baseline period.

   Behavioral Tasks: PRT, and IMT.

   Mobile Biobehavioral measures: ongoing data collection through continuous use of wearable sensors, peripherals, and EMA.

   NeuroBehavioral Unit: Will be "in-situ" (staying locally) during much of this time and spend one 24-hour period in the NBU (This will include NBU visit 3 of 8)

   Week 3-8: Following two weeks recovery, seen for initial DBS programming session for monopolar survey. The subject will be seen every 1-2 weeks for programming optimization.

   Repeat assessments:

   Clinician-administered: Vital Signs, MADRS, CGIS, YMRS, C-SSRS, HAM-A, MRTF, PRISE, Subject Reported: QIDS-SR, QOLS, SDS, BIS, ASRM, PANAS, MEQ, ISS.

   Neuropsychological Testing (Neuropsych): Likert-like scales assessing mood, anxiety and energy will be given before and after programming. Behavioral Tasks: PRT and IMT at month 1.

   Mobile Biobehavioral measures: ongoing data collection through continuous use of wearable sensors, peripherals, and EMA. Begin collection of LFPs to be synchronized other measures for offline analysis.

   Neurobehavioral Unit: One 24-hour stay in NBU. (NBU visits 4 and 5 out of 8 will occur during this time)

   Months 2-9: These will include once a month visits in order to optimize chronic DBS programming for efficacy and safety.

   Repeat assessments:

   Clinician-administered: Vital Signs, MADRS, CGIS, YMRS, C-SSRS, HAM-A, MRTF, PRISE,

   Subject Reported: QIDS-SR, QOLS, SDS, BIS, ASRM, PANAS, MEQ, ISS. Medical and Laboratory Testing: Repeat MEG, rsfMRI, at end-of-month 6.

   Neuropsychological Testing (Neuropsych): Repeat the neuropsych battery defined in the screening/baseline period.

   Behavioral Tasks: PRT, and IMT.

   Mobile Biobehavioral measures: ongoing data collection through continuous use of wearable sensors, peripherals, and EMA.

   NeuroBehavioral Unit: Will be "in-situ" (staying locally) during much of this time and spend one 24-hour period in the NBU.

   (This will be NBU visit 6 of 8)

   Month 9 visit: At this visit the team will determine if subject meets responder criteria

   Repeat Assessments:

   Clinician-administered: Vital Signs, MADRS, CGIS, YMRS, C-SSRS, HAM-A, MRTF, PRISE,

   Subject Reported: QIDS-SR, QOLS, SDS, BIS, ASRM, PANAS, MEQ, ISS.

   Medical and Laboratory Testing: Repeat MEG, rsfMRI.

   Neuropsychological Testing (Neuropsych): Repeat post-op baseline Neuropsych battery.

   Behavioral Tasks: PRT, and IMT at end-of-month 9.

   Mobile Biobehavioral measures: ongoing data collection through continuous use of wearable sensors, peripherals, EMA, and neural LFPs.

   NeuroBehavioral Unit: Will be "in-situ" (staying locally) during much of this time and spend one 24-hour period in the NBU.

   (This will be NBU visit 7 of 8)

   Months 9-12: Continuation of monthly visits for key clinical evaluations

   Repeat Assessments:

   Clinician-administered: Vital Signs, MADRS, CGIS, YMRS, C-SSRS, HAM-A, MRTF, PRISE,

   Subject Reported: QIDS-SR, QOLS, SDS, BIS, ASRM, PANAS, MEQ, ISS.

   Mobile Biobehavioral measures: ongoing data collection through continuous use of wearable sensors, peripherals, EMA, and neural LFPs.

   End Month 12: Begin 1 month withdrawal period. The DBS system will be turned off completely at some point during this gradual taper period. The study doctor will make the clinical decision whether to restart stimulation.

   Repeat Assessments:

   Clinician-administered: Vital Signs, MADRS, CGIS, YMRS, C-SSRS, HAM-A, MRTF, PRISE,

   Subject Reported: QIDS-SR, QOLS, SDS, BIS, ASRM, PANAS, MEQ, ISS.

   Medical and Laboratory Testing: Repeat MEG, rsfMRI,

   Behavioral Tasks: PRT, and IMT at end-of-month 12. NeuroBehavioral Unit: Will be "in-situ" (staying locally) during much of this time and spend one 24-hour period in the NBU.

   (This will be NBU visit 8 of 8)

   Months 13-20: The team and subject will make the clinical decision whether to reinstate or deactive DBS following discontinuation phase.

   Repeat Assessments:

   Clinician-administered: Vital Signs, MADRS, CGIS, YMRS, C-SSRS, HAM-A, MRTF, PRISE,

   Subject Reported: QIDS-SR, QOLS, SDS, BIS, ASRM, PANAS, MEQ, ISS.

   Month 20: Last set of formal study visits. All evaluations and labs will be repeated.

   Clinician-administered: Vital Signs, MADRS, CGIS, YMRS, C-SSRS, HAM-A, MRTF, PRISE,

   Subject Reported: QIDS-SR, QOLS, SDS, BIS, ASRM, PANAS, MEQ, ISS.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ages 22-64, inclusive
2. Diagnosis: Bipolar I disorder confirmed by SCID-5, currently in a major depressive episode (MDE).
3. Symptom Severity: MADRS score of ≥27 at Screening and pre-operative baseline visit. CGI-S > 4 and YMRS <12 at these visits.
4. Failure to respond or maintain a response to a minimum of four evidence-based interventions for bipolar depression in the patient's lifetime, including at least two FDA-approved medications (olanzapine/fluoxetine, quetiapine, lurasidone, cariprazine, lumateperone), or ECT, administered at adequate doses and duration (adequately defined by the Antidepressant Treatment History Form (ATHF-Short Form). During the current episode, the patient must have failed to respond or maintain a response to a minimum of two FDA-approved interventions for bipolar depression. In addition, the patient is required to be currently taking at least one evidence-based medication for bipolar disorder (e.g., lithium, either alone or in combination with an atypical antipsychotic such as quetiapine), unless no evidence-based medications for bipolar disorder are tolerated.
5. Initial mood episode occurred before the age of 40 - to minimize risk of enrolling patients with so atypical onset of initial mania/depression.
6. Must be on a stable dose of psychotropic medications for a minimum of four weeks prior to surgery.
7. Minimum score on the Montreal Cognitive Assessment (MoCA).
8. Able and willing to give informed consent and sign Treatment Contract that includes identification of a reliable informant.

Exclusion Criteria:

1. Lifetime history of a psychotic disorder (e.g., schizophrenia, schizoaffective disorder, and other psychotic disorders), or any history of psychotic symptoms when not in a bipolar mood episode.
2. Currently meets criteria for a manic or hypomanic episode or rapid cycling (4 or more mood episodes in the previous 12 months).
3. Any psychiatric disorder which is the primary focus of treatment within the past 12 months (with bipolar disorder as the secondary focus of treatment).
4. Alcohol/substance use disorder, moderate or severe, within the previous 12 months [excluding nicotine].
5. Intellectual disability or neurocognitive disorder.
6. Current major and/or unstable medical conditions. e.g., liver insufficiency, kidney insufficiency, cardiovascular problems [unstable arrhythmias, chronic heart failure, myocardial infarction (MI), cardiac pacemaker], systemic infections, cancer, active upper respiratory infections, endocrinopathies, and any major neurological disorder [e.g., seizure disorder, stroke, dementia, degenerative neurologic diseases, traumatic brain injury].
7. Any medical contraindication to surgery or condition that makes the patient, in the opinion of the surgeon, a poor candidate.
8. Female who is pregnant or breastfeeding or has plans to become pregnant in the next 24 months.
9. Any contraindication for MRI.
10. Patients with a clinically significant personality disorder, including risk for homicidal or aggressive behavior, which in the opinion of the investigator has a major impact on the patient's current psychiatric status and/or would preclude safe study participation.
11. Patients at serious and imminent risk of suicide and not suitable for an outpatient study, in the judgment of the investigators.
12. Participation in any investigational clinical trial within the preceding 30 days.
13. Current implanted stimulation devices including cardiac pacemakers, defibrillators, and neurostimulators [including deep brain and spinal cord stimulators].
14. Patients with no regular contact with at least one adult. Patients who are undomiciled are excluded.
15. Body mass index (BMI) less than 16 and greater than 40 kg/m2
16. Need for diathermy.
17. Unable to sign the informed consent for any reason.
18. Patients who are not under the care of a psychiatrist at Screening and throughout the duration of the study.

Ages: 22 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2029-05-30 (Estimated); Study Completion 2030-05-30 (Estimated)

PRIMARY OUTCOMES:
Utilizing the Montgomery-Asberg Depression Ratings Scale (MADRS) as a measurement of Efficacy | 20 months
  Efficacy: Primary outcome measure is a greater than or equal to 50% reduction on the Montgomery-Asberg Depression Ratings Scale (MADRS) at 9 months post-activation, compared to baseline score, which is obtained about 1 week pre-op. MADRS will evaluate Sadness, tension, Sleep, appetite, Concentration, and thoughts.
  This is a number scale with the higher number being a worse outcome
Utilizing the Patient-Rated Inventory of Side Effects (PRISE) assessment for adverse events/side effects | 20 months
  Adverse events will be elicited at each study visit using the PRISE, a standardized self-rating instrument, and confirmed by assessment of the study psychiatrist. Evaluation of manic episodes will be captured by clinical assessment to determine whether patients meet full or partial criteria for hypomanic, manic episodes, or mixed episodes. PRISE will be utilized to review Adverse Event criteria.The PRISE scale includes questions regarding subjects gastrointestinal status, heart status, skin status, nervous system status, eyes/ear status, genital/urinary status, sleep status, sexual functioning status, and "other" status with an area to specify any other concerns. This is a number scale with the higher number being a worse outcome
Evaluation of manic episodes utilizing the Young Mania Rating Scale (YMRS) | 20 months
  Evaluation of manic episodes will be captured by clinical assessment to determine whether patients meet full or partial criteria for hypomanic, manic episodes, or mixed episodes.This will be based on the Young Mania Rating Scale. This safety measures is administered at: screening, baseline, 1-week post-op, 2 weeks post-op (at activation visit), and then monthly for 20 months.
  The YMRS rating allows subjects to select from several categories to describe their level of energy. Some items include sleep, energy levels, sex drive, talkativeness, etc. This is a number scale with the higher number being a worse outcome
Evaluation of manic episodes utilizing the Altman Self-Rating Mania Scale (ASRM) | 20 months
  Evaluation of manic episodes will also be captured based on the self-report on the ASRM rating scale. This safety measures is administered at: screening, baseline, 1-week post-op, 2 weeks post-op (at activation visit), and then monthly for 20 months.
  The ASRMS rating allows subjects to select from several categories to describe their level of energy. Some items include sleep, energy levels, sex drive, talkativeness, etc. This is a number scale with the higher number being a worse outcome

SECONDARY OUTCOMES:
Durability of efficacy of the absence of recurring depressive episodes by utilizing the Montgomery-Asberg Depression Ratings Scale (MADRS) . | 20 months
  This secondary outcome measure is based on the durability of efficacy by utilizing the MADRS. Durability will be determined by the absence of recurrence of depressive episodes during the subsequent 9 months of observation (3 months stabilization, 6 months follow-up). Recurrence of a depressive episode is defined as a 25% increase of the MADRS over two consecutive monthly visits compared to score at 9 months post-activation = 6 "much worse" or 7 "very much worse" compared to the 9 months post-activation time point. The MADRS is completed by subjects indicating a 0-7. This is a number scale with the higher number being a worse outcome
Durability of efficacy of the absence of recurring depressive episodes by utilizing the Clinical Global Impressions Scale (CGI-S) | 20 months
  Another secondary outcome measure is durability of absence of recurring episodes will be evaluated by the CGI-S. This will be determined by the absence of recurrence of depressive episodes during the subsequent 9 months of observation (3 months stabilization, 6 months follow-up). Recurrence of a depressive episode is defined as a 25% increase of the CGI-S over two consecutive monthly visits compared to score at 9 months post-activation. CGI-S = 6 "much worse" or 7 "very much worse" compared to the 9 months post-activation time point. The CGI-s is completed by subjects indicating a 0-7. This is a number scale with the higher number being a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Goodman, MD, Principal Investigator — Baylor College of Medicine
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Baylor College of Medicine, Houston, Texas
  - Rice University, Houston, Texas
  - University of Washington, Seattle, Washington